CLINICAL TRIAL: NCT01114503
Title: A Randomised, Comparator Controlled, Two Part, Open-label Study to Evaluate the Safety, Tolerability and Pharmacodynamics of Multiple Doses of Otelixizumab in Patients With Thyroid Orbitopathy
Brief Title: A Safety and Tolerability Study of Otelixizumab in Thyroid Eye Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Clinical study in Graves' ophthalmopathy terminated until there is a better understanding of an efficacious dose with Otelixizumab from other clinical studies.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 112480; 2009-016747-19 (EudraCT Number)
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Graves Ophthalmopathy
Keywords: GSK2136525; Pharmacodynamics; Safety; Otelixizumab; Thyroid eye disease; Graves' ophthalmopathy; Repeat dose; Intravenous infusion; Tolerability; EUGOGO
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — otelixizumab; Methylprednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Part A (Experimental): Up to 4 cohorts of 5 patients receive dose rising treatments of otelixizumab
  Interventions: Drug: Otelixizumab - low dose; Drug: Otelixizumab - medium low dose; Drug: Otelixizumab - medium high dose; Drug: Otelixizumab - high dose
- Part B - Otelixizumab (Experimental): Parallel dosing group in Part B receive otelixizumab over 8 days at a dose decided upon results from Part A
  Interventions: Drug: Otelixizumab
- Part B - Methylprednisolone (Active Comparator): Parallel dosing group in Part B of weekly doses of methylprednisolone for 12 weeks
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Otelixizumab - low dose — 8 day dose rising intravenous infusions of a low dose of otelixizumab
  Arms: Part A
Drug: Otelixizumab - medium low dose — 8 day dose rising intravenous infusions of a medium low dose of otelixizumab
  Arms: Part A
Drug: Otelixizumab - medium high dose — 8 day dose rising intravenous infusions of a medium high dose of otelixizumab
  Arms: Part A
Drug: Otelixizumab - high dose — 8 day dose rising intravenous infusions of a high dose of otelixizumab
  Arms: Part A
Drug: Otelixizumab — 8 day dose rising intravenous infusions of otelixizumab administered at a dose decided upon results from Part A.
  Arms: Part B - Otelixizumab
Drug: Methylprednisolone — Weekly intravenous infusions of methylprednisolone administered as 500 mg per week for 6 weeks and then 250 mg per week for 6 weeks
  Arms: Part B - Methylprednisolone

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of otelixizumab in patients with Graves' ophthalmopathy (thyroid eye disease). There is currently no alternative therapy available for this condition other than treatment with steroids, or radiotherapy and surgery. The study also includes a comparison of the current steroid treatment, methylprednisolone, with the proposed new otelixizumab treatment.

DETAILED DESCRIPTION:
This is a study of otelixizumab, a monoclonal antibody (MAb) directed against the human lymphocyte antigen CD3 (a protein found on a certain type of white blood cell). This will be an open-label, comparator-controlled, two part study to evaluate the safety and tolerability of otelixizumab in patients with Graves' ophthalmopathy (GO). It will also look to see if otelixizumab affects GO and how it works compared to methylprednisolone (the standard treatment for active GO).

In Part A, between one and four groups of 5 patients will receive doses of otelixizumab administered over 8 days. The first dose level will provide a low cumulative dose, this low dose level has been safely administered in previous studies. Safety and clinical response data will be reviewed after 8 weeks, if no clinical response is seen and there are no safety concerns, the dose of otelixizumab will be increased and a new group of subjects will enter Part A. In subsequent groups cumulative medium low, medium high, and high doses of otelixizumab may be investigated. However if a clinical response is seen at the lowest dose the study will move directly to Part B.

In Part B, patients will receive either otelixizumab at the dose set from Part A, over 8 days (5 patients) or methylprednisolone weekly for 12 weeks (5 patients). All dosing will be by intravenous infusion. All participants will undergo long term safety evaluation for 48 months.

Key assessments include vital signs, 12-lead ECG, liver function tests, thyroid function, viral monitoring, monitoring of cortisol and ACTH levels, laboratory safety tests and adverse event (side effect) data. Assessment of GO severity will be evaluated using recommended assessments including clinical activity assessments and quality of life questionnaires. Measurements of exploratory biomarkers (proteins found naturally in the blood) are also included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 75 years of age inclusive
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 mIU/ml and estradiol <40 pg/ml (<140 pmol/L) is confirmatory].
* Child-bearing potential and agrees to use one of the agreed contraception methods listed in the protocol for an appropriate period of time to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception for at least 2 weeks prior to dosing and for at least 6 months after the last dose.
* Male subjects must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until at least 60 days after the last dose.
* Blood test of liver function within normal range
* Body mass index within 18.5 - 35 kg/m2 inclusive
* Capable of giving informed consent and agreement to comply with the study restrictions
* 12-lead ECG within normal limits
* fT4 blood levels within reference range for at least 2 months
* Active Graves' Ophthalmopathy (GO) with a Clinical Activity Score (CAS) of >/= 3 out of 7
* Moderately severe GO (as defined by EUGOGO guidelines)
* No previous immunosuppressive treatment for GO
* Subject is seropositive for EBV with <10,000 copies of EBV DNA per 10^6 lymphocytes (qPCR) or seronegative with no evidence of acute EBV infection (asymptomatic, negative EBV IgM and EBV viral load of <10,000 per 10^6 lymphocytes)
* The subject has no current or prior malignancy, other than non-melanoma skin cancer (subject must have had fewer than 5 occurrences of non-melanoma skin cancer, and the last occurrence must not be within 3 months of study entry)

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines
* Positive test for HIV antibody
* Positive test for syphilis
* History of regular alcohol consumption within 6 months of the study defined as:
* an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or
* an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females)
* Participation in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) or planning to take any investigational drug for the planned duration of study participation (6 months after the last dose of study drug)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Pregnant females as determined by positive (serum or urine) hCG test at screening or prior to dosing, or lactating females
* Currently receiving or has received corticosteroids or other immunosuppressive agents within the last 3 months
* Evidence of optic neuropathy and/or corneal breakdown
* Immunization with a vaccine within 30 days before the first dose of study drug or requires a vaccine within 30 days after the last dose of study drug
* A CD4+ lymphocyte count outside the range of 0.53 - 1.76 × 109/L during screening
* Significant systemic infection during the 6 weeks before the first dose of study drug
* Received a course of oral antibiotics within 2 weeks of dosing day one
* History of recurrent or chronic infection
* Subject has had a splenectomy
* Subjects with a screening chest X-ray suggestive of TB without documentation of adequate TB treatment
* Any major surgical procedure within the 8 weeks before signing the consent form, or planning to undergo any such surgery within the 3 months after the last dose of study drug
* Clinically significant cardiovascular and/or cerebrovascular disease
* Predisposition to thromboembolic disease, or thromboembolic event (excluding superficial) in past 12 months
* Uncontrolled medical conditions: Significant concurrent, uncontrolled medical condition including, but not limited to renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral psychiatric disease, or evidence of demyelinating disease
* A condition or situation that, in the investigator's judgment, is likely to cause the subject to be unable or unwilling to participate in study procedures or to complete all scheduled assessments
* Clinically significant abnormal laboratory values during the Screening period, other than those due to GO. Abnormal values are permitted if, upon re-test, the abnormality was resolved
* Unwillingness or inability to follow the procedures outlined in the protocol
* Mentally or legally incapacitated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-07-07 (Actual); Primary Completion 2012-08-29 (Actual); Study Completion 2012-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single center in United Kingdom from 23 June 2010 to 29 August 2012.
Pre-assignment Details: A total of 2 participants were randomized in cohort A1 of the study. The study was early terminated due to the need of better understanding of an efficacious dose with otelixizumab from other clinical studies.
Groups:
- Otelixizumab Cohort A1: Eligible participants received a total intravenous (IV) dose of otelixizumab 3.1 milligram (mg) for 8 days. The planned dosing regimen was 0.1 mg on Day 1, 0.2 mg on Day 2, 0.3 mg on Day 3, 0.5 mg on Day 4 to Day 8. The study medication was administered each day for 2 hours (h). The rate of infusion was 0.05 milligram per hour (mg/h) on Day 1, 0.1 mg/h on Day 2, 0.15 mg/h on Day 3, 0.25 mg/h on Day 4 to Day 8. At the start of each cohort in Part A, 2 participants acted as sentinel participants and complete dosing (Days 1-8) before further participants were dosed with otelixizumab. The first sentinel participants completed all of their dosing days and there was a minimum of 24 h elapse before the second sentinel participant started the dosing regimen. Further participants commenced dosing with otelixizumab once 24 h elapsed from the second sentinel participant receiving the final dose of otelixizumab on Day 8. Subsequent participants were dosed concurrently.
Period: Overall Study
Arm/Group | Otelixizumab Cohort A1
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Otelixizumab Cohort A1: Eligible participants received a IV dose of otelixizumab 3.1 mg for 8 days. The planned dosing regimen was 0.1 mg on Day 1, 0.2 mg on Day 2, 0.3 mg on Day 3, 0.5 mg on Day 4 to Day 8. The study medication was administered each day for 2 h. The rate of infusion was 0.05 mg/h on Day 1, 0.1 mg/h on Day 2, 0.15 mg/h on Day 3, 0.25 mg/h on Day 4 to Day 8. At the start of each cohort in Part A, 2 participants acted as sentinel participants and complete dosing (Days 1-8) before further participants were dosed with otelixizumab. The first sentinel participants completed all of their dosing days and there was a minimum of 24 h elapse before the second sentinel participant started the dosing regimen. Further participants commenced dosing with otelixizumab once 24 h elapsed from the second sentinel participant receiving the final dose of otelixizumab on Day 8. Subsequent participants were dosed concurrently.
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: Years] | 53.5 [53 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Adverse Event (AE), Serious Adverse Event (SAE), or Drug-related Adverse Event
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, associated with liver injury and impaired liver function defined as alanine aminotransferase >=3 x upper limit of normal (ULN), and total bilirubin >=2 x ULN or international normalized ratio >1.5. The classification as potentially drug-related was done based on the investigator's judgment.
Time Frame: Up to Month 24 (Long term follow-up)
Population: All Subjects Population included all participants who receive at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 2
Participants
  Any AE | 2
  Any SAE | 0
  Any drug-related (AE) | 2

2. Primary Outcome: Number of Participants With Laboratory Clinical Chemistry Abnormalities Meeting the Criteria for Potential Clinical Concern (PCC)
Description: The PCC range for clinical chemistry parameters included albumin, <30 gram per liter (g/L); calcium, low- < 2.0 millimole (mmol)/L: high->2.75 mmol/L; creatinine, high- > 1.3x ULN mmol/L or > 159 micromole (μmol)/L or > 44 μmol/L change from Baseline; glucose, low- < 3.0 mmol/L, high- > 9.0 0 mmol/L; magnesium, low- < 0.5 mmol/L, high- > 1.23 mmol/L, phosphorus, low- < 0.8 mmol/L, high- > 1.6 mmol/L; potassium, Low- < 3.0 mmol/L, high- > 5.5 mmol/L; sodium, low- < 130 mmol/L, high- > 150 mmol/L; bicarbonate, low- < 18 mmol/L, high- > 32 mmol/L; alanine aminotransferase, high->= 2x ULN, where the normal range was (NR) 0 - 39 international units (IU)/L; aspartate aminotransferase, high- >= 2x ULN, where NR was 0 - 39 IU/L; alkaline phosphatase, high- >= 1.5x ULN, where NR was 35 - 120 IU/L; total bilirubin- >= 1.5x ULN, where NR was 0 - 18 μmol/L.The assessments were done at Day 1 (pre dose), Day 8, Week 2-24 and Month 12 and 24.
Time Frame: Up to Month 24 (Long term follow-up)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 2
Participants | 0

3. Primary Outcome: Number of Participants With Laboratory Hematology Abnormalities Meeting the Criteria for PCC
Description: The PCC range for hematology parameters included white blood cell count, low- < 3 giga cells (GI)/L, high- > 20 GI/L; neutrophil count, low- < 1.5 GI/L; hemoglobin, low- > 25 g/L change from baseline, high- 180 g/L; hematocrit, low- > 0.075 L change from baseline, high- 0.54 L; platelet count, low- < 100 GI/L, high- >550 GI/L and lymphocytes, low < 0.8 GI/L. The assessments were done at Day 1 (pre dose), Day 8, Week 2-24, Month 12 and 24.
Time Frame: Upto Month 24 (Long term follow-up)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 2
Participants | 0

4. Primary Outcome: Number of Participants With Laboratory Urinalysis Abnormalities Meeting the Criteria for PCC
Description: The urinalysis parameters included pH, glucose, protein, blood and ketones by dipstic and microscopy (if urine dipstick was positive for blood or protein). The assessments were done at Day 1 (pre dose), Day 8, Week 2-24, Month 12 and 24.
Time Frame: Up to Month 24 (Long term follow-up)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 2
Participants | 0

5. Primary Outcome: Number of Participants With Thyroid Function Assessment, Hormone and Glucose Assay Abnormalities Meeting the Criteria for PCC
Description: The following laboratory parameters were analyzed: thyroid function assessment (thyroid stimulating hormone [TSH], thyroid peroxidase antibody, thyrotropin receptor antibodies (TSH-R-Abs) or TSH-binding inhibiting immunoglobulin (TBII), free thyroxine [fT4], free triiodothyronine [fT3]; hormone and glucose assays (cortisol, adrenocorticotrophic hormone [ACTH], insulin-like growth factor [IgF-1] and plasma glucose. Thyroid function tests were done at Day 1 (pre-dose) and Week 4-24. Hormone and glucose assays were done at Day 1 (pre-dose) and Week 2-24.
Time Frame: Up to Week 24
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 2
Participants | 0

6. Primary Outcome: Number of Participants With Vital Signs Abnormalities Meeting the Criteria for PCC
Description: Vital signs assessment included pulse rate, blood pressure, temperature and respiratory rate. Criteria for vital sign values meeting potential clinical concern included: supine pulse rate <40 or >110 beats per minute (bpm), >= 15 increase from baseline and >= 30 decrease from baseline; systolic blood pressure (SBP) < 85 and > 160 millimeters of mercury (mm Hg), >= 20 mmHg increase from baseline and >= 40 mmHg decrease from baseline; diastolic blood pressure (DBP) < 45 and > 100 mm Hg, >= 10 mmHg increase from baseline and >= 20 mmHg decrease from baseline.
Time Frame: Up to Month 24 (Long term follow-up)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 2
Participants | 0

7. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities Meeting the Criteria for PCC
Description: ECG parameters included pulse rate (PR) interval, QRS interval, QT interval, corrected QT interval using Bazett's formula (QTcB) and corrected QT interval using Fridericia's formula (QTcF). Criteria for ECG changes meeting potential clinical concern included: PR interval <110 and >220 milliseconds (msec); QRS interval <75 and >110 msec; QTc interval >480 to <= 500 msec, increase from baseline QTc >30 to <= 60 msec.
Time Frame: Screening (Day -35 to Day -1)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 2
Participants | 0

8. Primary Outcome: Number of Participants With an Epstein Barr Virus (EBV) Viral Load Abnormalities Meeting the Criteria for PCC
Description: The PCC range for EBV viral load was > 10,000 copies of deoxyribonucleic acid (DNA) per million lymphocytes. The assessments were done at Week 2, Week 4, Week 8 and Week 12.
Time Frame: Week 2 to Week 12
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 2
Participants | 0

9. Primary Outcome: Individual Absolute Circulating Peripheral T Lymphocytes (T-cells), CD4+ and CD8+ Subset Counts
Description: The lymphocyte subsets of T-cells, CD4+ and CD8+ cells were planned to be assessed at Day 1 (pre dose), Day 8 (pre dose), Week 2, Week 4, Week 8, Week 12 and Week 24. The absolute counts of the relevant lymphocyte subsets was to be determined by multiplying the percentages of the cell subsets with total lymphocyte counts. The percentages of relevant lymphocyte subsets was to be determined by flow cytometry. This endpoint was not analyzed due to the early termination of the study and since only 2 participants were recruited.
Time Frame: Up to Week 24
Population: All Subjects Population. No participants were available for analysis because of early termination of study.
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 0

10. Primary Outcome: Percentage of Circulating Peripheral T-cells, CD4+ and CD8+ Subset Counts
Description: The lymphocyte subsets of T-cells, CD4+ and CD8+ cells were planned to be assessed at Day 1 (pre dose), Day 8 (pre dose), Week 2, Week 4, Week 8, Week 12 and Week 24. The percentages of relevant lymphocyte subsets was to be determined by flow cytometry. This endpoint was not analyzed due to the early termination of the study and since only 2 participants were recruited.
Time Frame: Up to Week 24
Population: All Subjects Population. No participants were available for analysis because of early termination of study.
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 0

11. Primary Outcome: Assessment of CD3/T-cell Receptor (TCR) Complex Saturation and Modulation
Description: The assessment of CD3/TCR complex saturation and modulation was planned to be assessed on Day (1-8) pre dose, Week 2, Week 4, Week 8, Week 12 and Week 24. The extent of modulation was to be determined by the extent of TCR alpha beta (αβ) expression which was proportional to the combined levels of free CD3 sites and bound otelixizumab to CD4+ and CD8+ T cells. Bound levels of otelixizumab was planned to be determined by using flow cytometry method using an anti Immunoglobulin (Ig) antibody. The molecules of equivalent soluble fluorochrome (MESF) of the anti-Ig antibody was to be used to quantify the levels of bound otelixizumab present on T cells. Free otelixizumab binding sites (i.e., sites not occupied by otelixizumab administered to the participants) was to be detected by staining with fluorescein isothiocyanate (FITC) labelled otelixizumab. This endpoint was not analyzed due to the early termination of the study and since only 2 participants were recruited.
Time Frame: Up to Week 24
Population: All Subjects Population. No participants were available for analysis because of early termination of study.
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 0

12. Secondary Outcome: Change From Baseline for Individual Scores at Week 12 Incorporated in the European Group on Graves' Orbitopathy (EUGOGO) Assessment Including, Eyelid Swelling, Clinical Activity Score (CAS) Score, Proptosis, Lid Width and Diplopia
Description: The EUGOGO assessment of change was defined by improvement or deterioration of clinical scores. Improvement in EUGOGO was defined as improvement in two of the following measures in at least one eye, without deterioration in any of the same measures in both eyes: eyelid swelling according to color atlas evaluation, CAS by at least 2 points, proptosis by at least 2 millimeter (mm) by Hertel exophthalmometer, lid width by at least 2 mm, diplopia (disappearance or change in the degree) or improvement of >=8 degrees in motility unexplained by commensurate deterioration of motility of ipsilateral antagonists. Deterioration was defined by worsening by same quantity (as for improvement) of the same measures. Baseline was referred to assessment on Day 1 (pre dose). Change from Baseline was defined as post-Baseline value minus Baseline value. This endpoint was not analyzed due to the early termination of the study and since only 2 participants were recruited.
Time Frame: Baseline (Day 1, pre dose) and Week 12
Population: All Subjects Population. No participants were available for analysis because of early termination of study.
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 0

13. Secondary Outcome: Change From Baseline for Participant-reported Health Related Quality of Life (QoL) Questionnaires of Short Form 36 ( SF-36) and Graves Ophthalmopathy (GO) QoL
Description: Assessment of health related QoL was planned to be evaluated using the validated, disease specific, GO-QoL questionnaire and the SF-36 health survey questionnaire at Day 1 (pre dose) and Week 2- 24. Mean scores range from 0 (minimum) - 100 (maximum) with higher mean scores reflected better outcomes. Baseline was referred to assessment on Day 1 (pre dose). Change from Baseline was defined as post-Baseline value minus Baseline value. This endpoint was not analyzed due to the early termination of the study and since only 2 participants were recruited.
Time Frame: Baseline (Day 1, pre dose) to Week 24
Population: All Subjects Population. No participants were available for analysis because of early termination of study.
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 0

14. Secondary Outcome: Change From Baseline Measurement of Orbital Volume as Measured by Computed Tomography (CT) Scan
Description: The assessment of orbital volume measured by CT scan was planned to be assessed on Week 12 and Week 24. Baseline was referred to assessment at Screening. Change from Baseline was defined as post-Baseline value minus Baseline value. This endpoint was not analyzed due to the early termination of the study and since only 2 participants were recruited.
Time Frame: Baseline (Screening), Week 12 and Week 24
Population: All Subjects Population. No participants were available for analysis because of early termination of study.
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 0

15. Secondary Outcome: Assessment of Anti-otelixizumab Antibodies
Description: Anti-otelixizumab antibodies were planned to be assessed on Day 1 (pre dose), Day 8 (pre dose), Week 4-24 and Month 12. This endpoint was not analyzed due to the early termination of the study and since only 2 participants were recruited.
Time Frame: Up to Month 12
Population: All Subjects Population. No participants were available for analysis because of early termination of study.
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 0

16. Secondary Outcome: Assessment of Circulating Cytokines of Interleukin 6 (IL6), IL10, Interferon Gamma (IFNγ) and Tumor Necrosis Factor Alpha (TNFα) up to 2 Weeks
Description: Assessment of circulating cytokines of IL6, IL10, IFNγ and TNFα was planned to be assessed on Day 1-8 (pre dose) and Week 12. This endpoint was not analyzed due to the early termination of the study and since only 2 participants were recruited.
Time Frame: Up to Week 2
Population: All Subjects Population. No participants were available for analysis because of early termination of study.
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 0

17. Secondary Outcome: Assessment of Exploratory Biomarkers
Description: The exploratory biomarkers were planned to be assessed on Day 1 (pre dose), Week 4, Week 12 and Week 24. It included assessment of peripheral blood mononuclear cells (PBMC) markers, suppression assays for the measure of effector cell proliferation, quantification of effector memory T-cells subsets, autoreactivity assays using cytokine production of supernatants and CFSE dilution, cytokine production by in-vitro stimulated T-cells, circulating serum biomarkers and may include subsequently discovered biomarkers of the biological response associated with GO or medically related conditions and/or the action of otelixizumab. This endpoint was not analyzed due to the early termination of the study and since only 2 participants were recruited.
Time Frame: Up to Week 24
Population: All Subjects Population. No participants were available for analysis because of early termination of study.
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 0

18. Secondary Outcome: Assessment of Exploratory Biomarkers of Ribonucleic Acid (RNA) Transcription Analysis of Peripheral Blood
Description: The exploratory biomarkers of RNA transcription analysis of peripheral blood was planned to be assessed on Day 1(pre dose), Week 4 and Week 24. The assessment was to be done using microarray and RNA expression using quantitative reverse transcription polymerase chain reaction (RT-PCR). This endpoint was not analyzed due to the early termination of the study and since only 2 participants were recruited.
Time Frame: Up to Week 24
Population: All Subjects Population. No participants were available for analysis because of early termination of study.
Arm/Group | Otelixizumab Cohort A1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AE's and SAE's were recorded from Day 1 up to Month 24
Description: All Subjects Population was used.
Arm/Group | Otelixizumab Cohort A1
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Otelixizumab Cohort A1 (N=2)
Headache (Nervous system disorders) | 2
Foreign body sensation in eyes (Eye disorders) | 2
Hot Flush (Vascular disorders) | 1
Eye Pain (Eye disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to the need of better understanding of an efficacious dose with otelixizumab from other clinical studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.